CLINICAL TRIAL: NCT01657838
Title: A Phase 1, Randomized, Open-Label, Two-Arm, Parallel Group Study of the Effect of Ketoconazole at Steady State on the Pharmacokinetics of a Single Dose of Isavuconazole in Healthy Adult Subjects
Brief Title: Drug Interaction Study of the Effect of Ketoconazole at Steady State on the Pharmacokinetics of a Single Dose of Isavuconazole in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 9766-CL-0040
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Ketoconazole; Healthy Adult Volunteers
Keywords: Isavuconazole; Ketoconazole; Healthy Volunteers; BAL8557; BAL4815
MeSH Terms: interventions — isavuconazole; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: isavuconazole only (Experimental): Single dose of isavuconazole on Day 1
  Interventions: Drug: Isavuconazole
- Arm 2: isavuconazole + ketoconazole (Experimental): Single dose of isavuconazole on Day 4 and ketoconazole twice daily (BID) for 24 days
  Interventions: Drug: Isavuconazole; Drug: Ketoconazole

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL4815; BAL8557
Drug: Ketoconazole — oral
  Arms: Arm 2: isavuconazole + ketoconazole

SUMMARY:
The purpose of this study is to assess the effect of ketoconazole at steady state on the pharmacokinetics of a single dose of isavuconazole in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and total bilirubin must not be above the normal range
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy during the study period

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a positive result for hepatitis C antibodies or hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of occasionally use of ibuprofen
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for isavuconazole (in plasma): AUClast , Cmax | Day 1 (Arm 1) and Day 4 (Arm 2): predose and 0.5, 1, 2, 4, 6, 8, 10, 12, 20, 24, 36, 48, 72, 96,120,144,168,192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480 and 504 hours post-dose
  Area under the concentration-time curve from time of dosing to the last quantifiable concentration (AUClast) and maximum concentration (Cmax)

SECONDARY OUTCOMES:
PK profile for isavuconazole (in plasma): AUCinf, tmax, CL/F, Vz/F, and t1/2 | Day 1(Arm 1) and Day 4 (Arm 2): predose and 0.5, 1, 2, 4, 6, 8, 10, 12, 20, 24, 36, 48, 72, 96,120,144,168,192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480 and 504 hours post-dose
  Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf), Time to attain Cmax (tmax), apparent body clearance after oral dosing (CL/F), apparent volume of distribution (Vz/F), and apparent terminal elimination half-life (t1/2)
PK for ketoconazole (in plasma): trough concentration (Ctrough) | Day 2 (Arm 2): predose
PK profile for ketoconazole (in plasma): AUCtau, Cmax, and tmax | Days 3 and 4: predose and 0.5,1, 2, 4, 6, 8,12 and 24 hours post-dose
  AUC during time interval between consecutive dosing (AUCtau)
Safety assessed by recording of adverse events, clinical laboratory evaluation, electrocardiograms (ECGs) and vital signs | Day 1 through Day 25 (± 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States